CLINICAL TRIAL: NCT01380938
Title: RCT Comparing Different Ribavirin Dosages and Durations of Treatment in Combination With Peginterferon in HCV Genotypes 2 and 3 (WRITE)
Brief Title: Different Ribavirin Dosages and Different Duration of Treatment in Combination With PegInterferon in Patients With Genotype 2 and 3 (WRITE)
Acronym: WRITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: Casa di Cura Mater Dei (Unknown); IRCCS L. Spallanzani (Unknown); Ospedale Francesco Ferrari (Other); Azienda Ospedaliero Universitaria di Sassari (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Arcispedale S. Anna, Ferrara (Unknown); Azienda Ospedaliero-Universitaria, Catania (Unknown); Ospedale di Venosa (Unknown); Ospedale Monsignor R. Dimiccoli, Barletta (Other); IRCCS De Bellis, Castellana (Unknown); USL Napoli 1 (Unknown); Ospedale San Giuseppe Moscati, Avellino (Unknown); Cardarelli Hospital (Other); Ospedale Civile Vittorio Emanuele II, Bisceglie (Unknown); Azienda Ospedaliero-Universitaria Careggi (Other); Azienda Ospedaliera V. Cervello (Other); Ospedale Civile Spirito Santo (Other); Ospedale di Canosa di Puglia (Unknown); University of Palermo (Other); San Camillo Hospital, Rome (Other); Campus Bio-Medico University (Other); Ospedale Sandro Pertini, Roma (Other); Ospedali Riuniti di Foggia (Other); Ospedale SS. Annunziata, Taranto (Unknown); Ospedale di Mottola (Unknown); Ospedale Santa Caterina Novella, Galatina (Unknown); University of Florence (Other); Ospedale Valduce, Como (Unknown); University of Bari (Other); Azienda Ospedaliera, Siracusa (Unknown); Azienda Ospedaliera, Lucca (Unknown)
Responsible Party: Principal Investigator, Alessandra Mangia, MD, Casa Sollievo della Sofferenza IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPAT-01-2010
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Chronic Hepatitis
Keywords: genotypes 2 and 3; combination treatment; individualized treatment
MeSH Terms: conditions — Hepatitis, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm C. Standard duration (No Intervention): Patients will be randomly assigned in 3:3:1 ratio to three treatment arms. In the standard treatment group (Arm C), patients will be treated for 24 weeks independently of the HCV RNA status at week 4 with Peginterferon alpha-2a at a dose of 180 mcg weekly in combination with oral ribavirin administered at a dosage of 800 mg/day.
  Patients enrolled in Arm C will be treated for standard 24 weeks duration of treatment.
- Arm A (Experimental): Patients enrolled in Arm A will receive Peginterferon alpha-2a at a dosage of 180 mcg weekly in combination with oral ribavirin administered at a dosage of 1000 mg/day for patients with a body weight < 75 kg or 1200 mg/day for those with a body weight > 75 kg.
  Patients with week 4 viral clearance (labelled as rapid virological responders, RVR) will be allocated to 12 week treatment duration (Arm A), whereas those without RVR will be treated for 24 weeks (Arm A)
  Interventions: Drug: Peginterferon alpha-2a + Ribavirin
- Arm B (Experimental): Patients enrolled in Arm B will receive Peginterferon alpha-2a at a dosage of 180 mcg weekly in combination with oral ribavirin administered at a dosage of 800 mg/day.
  Patients with week 4 viral clearance (labelled as rapid virological responders, RVR) will be allocated to 12 week treatment duration (Arm B), whereas those without RVR will be treated for 48 weeks (Arm B)
  Interventions: Drug: Peginterferon alpha-2a + Ribavirin

INTERVENTIONS:
Drug: Peginterferon alpha-2a + Ribavirin — Administration of ribavirin at a dosage of 1000 or 1200 mg per day based on body weight < or > 75 kg for 24 weeks (Arm A).
  Treatment duration of 48 weeks with standard fixed dose of ribavirin (800 mg/day) (Arm B).
  These schedules will be compared with diagram of standard therapy with 800 mg daily of ribavirin for 24 weeks (Arm C)
  Other Names: Peginterferon alpha-2a (40 kD) PEGASYS; Copegus or Rebetol, Ribavirin Teva
  Arms: Arm A; Arm B

SUMMARY:
WRITE study aim at identifying the effectiveness of an innovative individualized schedule of treatment as compared to standard regimen in patients with chronic HCV genotype 2 and 3.

DETAILED DESCRIPTION:
The investigators are going to compare weight-based dosages of ribavirin, in combination with Peginterferon alpha-2a, with standard fixed dosages of 800 mg. Patients will be evaluated at week 4 with an assay of sensitivity of 15 IU/ml. Patients with week 4 response will discontinue treatment at week 12 in both arms. Patients with HCV RNA still detectable at week 4 and receiving 1000-1200 mg of ribavirin in arm A will discontinue treatment at week 24, whereas patients with HCV RNA still detectable at week 4 and receiving 800 mg of ribavirin in arm B will be treated till week 48.

A standard treatment arm (C) including patients treated for 24 weeks with Peginterferon alpha-2a and fixed 800 mg ribavirin dosage will be used as control arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C virus (HCV) infection (both HCVAb and HCV RNA positive)
* Patients with HCV genotype 2 or 3
* Age 18-70 years
* Naïve patients or previously treated only with standard interferon monotherapy
* Female patients of childbearing age who agree to avoid pregnancy during the period of treatment and 24 weeks after the end of treatment

Exclusion Criteria:

* Previous treatment with ribavirin
* Cirrhosis (CHILD PUGH B and C)
* Evidence of Hepatocellular carcinoma
* Pregnancy
* Retinopathy class I or II
* Alcohol consumption > 40 gr/day
* Chronic cardiac or respiratory diseases
* HIV or HBsAg or HDV positivity
* Hemoglobin < 8.5 gr/dL
* WBC < 3.500/mm3
* PLT < 80.000/mm3

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Sustained virological Response (SVR) | 6 months after the end of treatment
  The primary measure of efficacy will be HCV RNA not detectable in serum samples 24 weeks after the end of therapy (SVR).

SECONDARY OUTCOMES:
Rapid virological response (RVR) | On treatment week 4
  proportion of patients with undetectable HCV RNA 4 weeks after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Mangia, MD, Study Director — IRCCS "Casa Sollievo della Sofferenza"
Locations (35):
- Italy (35):
  - Infectious Diseases Unit, Avellino
  - Clinical Medicine Unit "Mater Dei", Bari
  - Università di Bari, Bari
  - Medicine Unit, Barletta
  - Infectious Diseases Unit "V. Emanuele", Bisceglie
  - Medicine Unit, Canosa di Puglia
  - Hepatology Unit, Casarano
  - IRCCS "De Bellis", Castellana Grotte
  - Hepatology Unit, Catania
  - Infectious Diseases Unit, Catania
  - Gastroenterology Unit, Como
  - Gastroenterology Unit Arcispedale "S. Anna", Ferrara
  - Gastroenterology Unit, Florence
  - Internal Medicine University of Firenze, Florence
  - Gastroenterology Unit, Foggia
  - Infectious Diseases, Foggia
  - Gastroenterology Unit, Galatina
  - Infectious Diseases, Lucca
  - Gastroenterology Unit, Mottola
  - Gastroenterology Unit "Cardarelli", Napoli
  - USL Napoli 1, Napoli
  - Hospital "V. Cervello", Palermo
  - Medical Clinic University of Palermo, Palermo
  - Infectious Diseases Unit IRCCS "San Matteo", Pavia
  - Campus Biomedico University, Roma
  - Hepatology Unit "S. Pertini", Roma
  - Hepatology Unit "san Camillo", Roma
  - Ospedale "Villa Betania", Roma
  - IRCCS "L. Spallanzani", Rome
  - IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo
  - Infectious Diseases Unit Ospedale Civile, Sassari
  - Medicine Unit, Sassari
  - Infectious Diseases, Syracuse
  - SS. Annunziata, Taranto
  - Medicine Unit, Venosa

REFERENCES:
- [Background] Mangia A, Dalgard O, Minerva N, Verbaan H, Bacca D, Ring-Larsen H, Copetti M, Carretta V, Piazzolla V, Cozzolongo R, Mottola L, Andriulli A. Ribavirin dosage in patients with HCV genotypes 2 and 3 who completed short therapy with peg-interferon alpha-2b and ribavirin. Aliment Pharmacol Ther. 2010 Jun;31(12):1346-53. doi: 10.1111/j.1365-2036.2010.04290.x. Epub 2010 Mar 8. PMID 20222909
- [Background] Mangia A, Minerva N, Bacca D, Cozzolongo R, Agostinacchio E, Sogari F, Scotto G, Vinelli F, Ricci GL, Romano M, Carretta V, Petruzzellis D, Andriulli A. Determinants of relapse after a short (12 weeks) course of antiviral therapy and re-treatment efficacy of a prolonged course in patients with chronic hepatitis C virus genotype 2 or 3 infection. Hepatology. 2009 Feb;49(2):358-63. doi: 10.1002/hep.22679. PMID 19072829
- [Background] Andriulli A, Mangia A, Iacobellis A, Ippolito A, Leandro G, Zeuzem S. Meta-analysis: the outcome of anti-viral therapy in HCV genotype 2 and genotype 3 infected patients with chronic hepatitis. Aliment Pharmacol Ther. 2008 Aug 15;28(4):397-404. doi: 10.1111/j.1365-2036.2008.03763.x. Epub 2008 Jun 11. PMID 18549461
- [Background] Mangia A, Santoro R, Minerva N, Ricci GL, Carretta V, Persico M, Vinelli F, Scotto G, Bacca D, Annese M, Romano M, Zechini F, Sogari F, Spirito F, Andriulli A. Peginterferon alfa-2b and ribavirin for 12 vs. 24 weeks in HCV genotype 2 or 3. N Engl J Med. 2005 Jun 23;352(25):2609-17. doi: 10.1056/NEJMoa042608. PMID 15972867